CLINICAL TRIAL: NCT01463956
Title: Pilot Study on the Efficacy of Pegylated Interferon-Ribavirin-Boceprevir Triple Therapy in Patients Infected With Genotype 1 HCV With Cirrhosis and Awaiting Liver Transplantation (ANRS HC 29 BOCEPRETRANSPLANT)
Brief Title: Efficacy of PegInterferon-Ribavirin-Boceprevir Therapy in Patients Infected With G1 HCV With Cirrhosis, Awaiting Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011- 001089 -17
Record Dates: First submitted 2011-10-14; First posted 2011-11-02 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: HCV Infection; Liver Cirrhosis, Experimental
Keywords: Boceprevir; HCV infection; Antiviral therapy; Liver transplantation
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis, Experimental | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boceprevir, Pegylated interferon and Ribavirin (Experimental): * Lead-in phase (4 week): Pegylated interferon + Ribavirin
  * Triple therapy regimen for 44 weeks :Boceprevir + Pegylated interferon + Ribavirin
  * Pegylated interferon + Ribavirin therapy until transplantation (less or equal to 24 weeks)
  Interventions: Drug: Boceprevir; Biological: Peg-Interferon α-2b or Peg-Interferon α-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — Boceprevir 200 mg capsules at 2400mg/day (800mg 3 times a day) from week 4 until week 48 or until liver transplant (can be performed from week 16)
Biological: Peg-Interferon α-2b or Peg-Interferon α-2a — Peg-Interferon α-2b by subcutaneous injection, 1.5µg/kg/week, from day 0 until week 48 or until liver transplantation, or Peg-Interferon α-2a by subcutaneous injection, 180 µg, once weekly, from day 0 until week 48 or until liver transplantation
  Other Names: PegIntron; PEG
Drug: Ribavirin — Ribavirin: capsules 200 mg (weight-based daily dose: <65kg, 800 mg; 65-80kg, 1000mg; 81-105kg: 1200mg; >105kg: 1400mg), from day 0 until week 48 or until liver transplantation or, Ribavirin: Tablet Oral, weight-based dose, 1000 mg for subjects weighing below 75 kg or 1200 mg for subjects weighing equal or over75 kg, once daily, from day 0 until week 48 or until liver transplantation

SUMMARY:
Evaluation of efficacy of triple therapy with pegylated interferon, ribavirin, and boceprevir in patients with genotype 1 chronic hepatitis C, who are treatment-naive, have relapsed, or are non-responders with cirrhosis and awaiting liver transplantation, with a MELD score less than or equal to 18

DETAILED DESCRIPTION:
Evaluation of sustained virological response defined as the proportion of patients with undetectable hepatitis C virus RNA 24 weeks after discontinuation of therapy and/or after liver transplantation in patients with genotype 1, who are treatment-naive, have relapsed, or are non-responders with cirrhosis and awaiting liver transplantation, with a MELD score less than or equal to 18

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years and older
* Chronic infection with hepatitis C virus proven with positive PCR for more than 6 months
* Viral genotype 1
* Cirrhosis while awaiting liver transplantation
* MELD score < or equal to 18
* With or without hepatocellular carcinoma
* Naive to antiviral C treatment
* Failure on a previous treatment. Failure is defined as the persistence of detectable HCV RNA. The previous HCV failure treatment profile must be able to be documented according to the following terminology:- Relapsing patient: HCV RNA undetectable at the end of treatment, becoming detectable again after the discontinuation of treatment- Breakthrough: increase of viremia of 1 log or more during the treatment - Non-responding patient with partial response: HCV RNA detectable at W24 without ever having been undetectable and with a decrease in HCV RNA ≥ 2 log at W12 - Non-responding patient with nul response: decrease in HCV RNA < 2 log at W12
* No need for prior treatment wash-out
* Negative pregnancy test in women of child-bearing age
* Double method of contraception in men and women of child-bearing age during the entire duration of treatment and the 6 months following its discontinuation
* Free, informed, and written consent (signed on the day of pre-enrollment at the latest and before all exams required by the study)
* Person enrolled in or a beneficiary of a social security/Universal Health Insurance Coverage
* Inclusion approved by the Decision Support Committee

Exclusion Criteria:

* Previous HCV treatment with boceprevir or telaprevir
* Alcohol consumption > 40 g/day
* Toxicomania constituting a barrier for starting therapy according to the opinion of the investigator. Patients included in a methadone or buprenorphine replacement program may be enrolled
* MELD > 18
* Non controlled sepsis
* Platelets < 50,000/mm3
* Neutrophil granulocyte levels < 1000/mm3
* Creatinine clearance < 50 mL/min (MDRD)
* Hb < 10 g/dL
* Uncontrolled psychiatric problems
* Contraindications to boceprevir
* Contraindication to interferon or ribavirin
* Subject with major complications of cirrhosis
* HIV coinfection
* HBV coinfection (unless this is treated effectively with analogues, as proven by undetectable viremia for at least 12 months)
* Other infectious disease underway
* Neoplastic disease other than hepatocellular carcinoma during the previous year, or neoplastic disease for which the prognosis is less than 3 years
* Treatment with immunosuppressors (including corticosteroids), antivirals other than those for the study, except aciclovir
* Consumption of St. John's wort
* Associated treatments including a molecule or substance that could interfere with the pharmacokinetic characteristics of boceprevir
* History of a lactose allergy
* Person participating in another study including an exclusion period that is still underway during pre-enrollment
* So-called vulnerable populations (minors, people under guardianship or protection, or a private individual under protection from making legal or administrative decisions)
* Pregnancy, breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-01-06; Primary Completion 2014-06 (Actual); Study Completion 2015-01-22 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) Rate | Week 24 after the discontinuation of antiviral C treatment and at the time of liver transplantation or at the time of liver transplantation
  Evaluation of sustained virologic response to antiviral C treatment depends of time of liver transplantation that can be performed between week 16 and week 96 of the trial:
  * If the liver transplant is realized after the discontinuation of antiviral C treatment,sustained virologic response should be evaluated 6 months after the discontinuation of antiviral C treatment and at the time of liver transplantation.
  * If the liver transplant is realized before the discontinuation of antiviral C treatment,sustained virologic response should be evaluated at the time of liver transplantation.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | From week 0 to week 144
  Information on adverse events will be collected by the investigator during medical visits and reported in the CRF. Adverse events will be classified as: a) Flu-like symptoms b) Musculoskeletal symptoms c) Neurologic symptoms d) Psychiatric symptoms e) Constitutional symptoms
Perceived symptoms | at day 0, week 24, week 48 and every 24 week up liver transplant - post liver transplant: day 0, week 24 and week 48
  Information on symptoms as perceived by the patients will be collected through self-administered questionnaires.
Compliance rate. | week 12, week 24, week 36, week 48, week 72 - after Liver transplant:Day 0
  Treatment compliance will be assesses through a self-administered questionnaire reporting the number of medication doses prescribed and taken by the participants
SVR prognosis factors | Week-4 up week 144
  Participants with undetectable plasma HCV-RNA 24 weeks after treatment cessation and/or liver transplantation will be considered as SVR. Factors potentially associated with SVR will be studied through a logistic regression analysis. These factors include demographical (age, gender), virological (baseline viral load), clinical (disease severity measured by MELD score) and genetic factors (IL28B polymorphism: TT, CT, or CC)
The predictive value of on-treatment HCV RNA on SVR | During weeks 1, 4, 5, 6, 7, 8, 12, 16, 20, and 24 (before transplantation)
  Quantitative assessment of HCV RNA during treatment will be performed at weeks 1, 4, 5, 6, 7, 8, 12, 16, 20, and 24 and correlated to SVR
The percentage of virologic failure | week 4 and week 48
  Virological failure is defined as an increase of HCV RNA of at least 1 log IU/mL during treatment, or by the reappearance of positive viremia during treatment, after an initial negative result
The percentage of relapse after transplantation | Between week 16 and week 144
  Virological relapse is characterized by an HCV RNA negative at the end of treatment but becoming detectable after cessation of therapy. The proportion of patients with virological relapse will be determined
Boceprevir resistant mutations | From week 5 to week 48 or after week 48
  The proportion of patients with emergence of resistant mutations to boceprevir in case of detectable viral load during treatment (from W5) and after the discontinuation of treatment in the event of virologic failure will be assessed
Resistant mutations in plasma and liver samples (both explanted liver and graft) | Week 16 up to week 96
Sepsis according to Systemic Inflammatory Response System (SIRS) Criteria | From day 0 to week 72
Cirrhosis impairment | From day 0 to week 72
  Cirrhosis impairment will be assessed by studying:
  * the mean variation of MELD score between baseline and end of therapy
  * the proportion of patients with a MELD score increased by at least 3 points (in case of baseline MELD>15) or 5 points (in case of baseline MELD<15)
Survival after transplantation | Week 16 up to week 96
Survival rate within one year after liver transplantation | week 64 up to week 144
The mean time elapsed between registration on the transplantation list and the date of transplantation | Week16 up to week 96
Measurement of the residual plasma concentration (Cres) of ribavirin | at Week 4 and Week 8
Area Under the Plasma Concentration Time Curve (AUC) From 0-8h of Boceprevir | At week 16 and at week 24 and if the MELD score has changed by more than three points
Maximum Plasma Concentration (Cmax) of Boceprevir | At week 16 and at week 24 and if the MELD score has changed by more than three points
Time of Maximum Plasma Concentration (Tmax) of Boceprevir | At week 16 and at week 24 and if the MELD score has changed by more than three points
Minimum Plasma Concentration (Cmin) of Boceprevir | At week 16 and at week 24 and if the MELD score has changed by more than three points
Correlation study between the presence of an elevated level of IP-10 during triple therapy and the absence of sustained virologic response | From week 4 to week 48
  Plasma aliquots will be performed in all patients of the trial at day 0 before liver transplant and day 0 post liver transplant to measure IP10. Evaluation will be performed at the end of the trial for all patients recruited. The association between IP-10 level and SVR will be assessed
Histological severity of HCV recurrence after liver transplantation | At week 20 up to week 100, at week 40 up to week 120, at week 64 up to week 144
  Histological severity will be assessed by the METAVIR score at 1 month (if early recurrence), at 6 months, 1 year after transplantation in case of non-response/relapse before transplantation .
  Liver transplantation can be performed between week 16 and week 96
Insulin Resistance (HOMA-IR) | At baseline, week 48 and at the last follow-up visit
Virological Response in participants with and without Insulin Resistance | At week 4, 8, 16, 28 and 48 during therapy
Relationship between the presence of a polymorphism in the IL28B gene (donor and recipient) and SVR | After week 144
  Whole blood aliquots (DNA bank) will be performed at the Day 0 visit to measure IL28B polymorphism. Evaluation will be performed at the end of the trial for all patients recruited. The SVR rate will be compared between the different IL28B phenotypes (CC, CT and TT).
Relationship between the presence of a polymorphism to the ITPA gene and the onset of hemolytic anemia | After week 144
  Whole blood aliquots (DNA bank) will be performed at the Day 0 visit for ITPA gene measure. Evaluation will be performed at the end of the trial for all patients recruited. The proportion of patients with occurrence of hemolytic anemia will be compared according to the ITPA polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Didier Samuel, Pr, Principal Investigator — Hepatobiliary Center of Paul Brousse Hospital. France
Locations (19):
- France (19):
  - Haut-Lévêque Hospital, Bordeaux
  - Beaujon Hospital, Clichy
  - Henri Mondor Hospital, Créteil
  - A Michallon Hospital, Grenoble
  - Claude Huriez hospital, Lille
  - La Croix-Rousse, Lyon
  - La Conception Hospital, Marseille
  - Saint-Eloi Hospital, Montpellier
  - Archet Hospital, Nice
  - La Pitié Salpétrière Hospital, Paris
  - Cochin Hospital, Paris
  - Staint Antoine Hospital, Paris
  - Pontchaillou Hospital, Rennes
  - Civil Hospital, Strasbourg
  - Purpan Hospital Médecine interne, Toulouse
  - Purpan Hospital, Toulouse
  - Trousseau Hospital, Tours
  - Nancy Hospital, Vandœuvre-lès-Nancy
  - Paul Brousse Hospital, Villejuif